CLINICAL TRIAL: NCT04190082
Title: The Effect of Bispectral Index Monitoring on the Speed of Recovery From Deep Propofol Sedation in Children With Cerebral Palsy - A Randomized Controlled Trial
Brief Title: The Effect of Bispectral Index Monitoring on Recovery From Deep Sedation
Status: Terminated | Type: Observational
Why Stopped: No more participants enrolled.
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sung Mee Jung, Professor, Yeungnam University College of Medicine
Other Study IDs: YUMC-2019-11-001
Record Dates: First submitted 2019-12-04; First posted 2019-12-09 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Botulinum toxin; Bispectral index monitor; Deep sedation; Recovery
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Control: Group who maintains deep sedation using the University of Michigan sedation scale (UMSS) score.
- Group BIS: Group who maintain deep sedation using Bispectral Index (BIS) score.

SUMMARY:
The purpose of this study was to compare BIS (bispectral index) monitoring and clinical sedation scale assessment on the recovery time and propofol usage from deep propofol sedation in children with cerebral palsy who received botulinum toxin injection.

DETAILED DESCRIPTION:
After arrival in the preoperative holding area, children were randomly allocated into two groups using a computer-generated random assignment scheme. Five minutes before propofol sedation, remifentanil is administered intravenously at 0.025 μg / kg / min for analgesic effect and continued throughout the sedation process until just before the end of the procedure. Five minutes after remifentanil administration, 2 mg / kg of propofol mixed with 1 mg / kg of lidocaine was administered over 30 seconds, followed by continuous infusion at 100 μg / kg / min. Group C is monitored using UMSS(University of Michigan Sedation Scale) scores every three minutes, and group B is monitored using BIS score until deep sedation. Deep sedation is defined based on UMSS score of 3-4 and BIS score of 65 ± 5. If the sedation score is determined to have reached a deep sedation, a botulinum toxin injection is given by a practitioner blind to how to assess the depth of sedation. Independent investigator who is blind to group assignement assesses the oxygen saturation, respiration, and blood pressure, recovery time from sedation, and adverse events during and after sedation.

ELIGIBILITY:
Inclusion Criteria:

* 3-12 years old children with spastic cerebral palsy receiving botulinum toxin injection with deep sedation
* American Society of Anesthesiologists Physical Status 1-2

Exclusion Criteria:

* Body mass index > 30 kg/m2
* unstable heart disease
* Anticipated difficult airway including congenital facial or airway anomaly
* Recent upper respiratory tract infection ( < 2 weeks)
* Gastroesophageal reflux
* Allergy history to propofol, remifentanil or any drug used during procedure

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with spastic cerebral palsy primary care clinic (rehabilitation)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
recovery | Immediately after discontinuation of propofol infusion used for botulinum toxin injection
  Time taken to recover based on the Physiological CBD score (>12) from deep sedation

SECONDARY OUTCOMES:
Propofol dose | Immediately after discontinuation of propofol infusion used for botulinum toxin injection
  Amount of propofol to maintain deep sedation for botulinum toxin injection

CONTACTS AND LOCATIONS:
Overall Officials: Sung Mee Jung, MD,PhD, Principal Investigator — Yeungnam University Hospital
Locations (1):
- Location Yeungnam University Hospita, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share our data

REFERENCES:
- [Result] Choudhry DK, Brenn BR. Bispectral index monitoring: a comparison between normal children and children with quadriplegic cerebral palsy. Anesth Analg. 2002 Dec;95(6):1582-5, table of contents. doi: 10.1097/00000539-200212000-00020. PMID 12456420
- [Result] Malviya S, Voepel-Lewis T, Tait AR. A comparison of observational and objective measures to differentiate depth of sedation in children from birth to 18 years of age. Anesth Analg. 2006 Feb;102(2):389-94. doi: 10.1213/01.ANE.0000184045.01780.73. PMID 16428530
- [Result] Saricaoglu F, Celebi N, Celik M, Aypar U. The evaluation of propofol dosage for anesthesia induction in children with cerebral palsy with bispectral index (BIS) monitoring. Paediatr Anaesth. 2005 Dec;15(12):1048-52. doi: 10.1111/j.1460-9592.2005.01658.x. PMID 16324022